CLINICAL TRIAL: NCT01213667
Title: Pharmacogenetics in Anti-VEGF Treatment Non-responders Suffering Exudative Age-related Macular Degeneration (AMD): Genetic Correlations and Intraocular Cytokine Concentrations
Brief Title: Genetics in Non-response to Anti-VEGF Treatment in Exudative AMD
Acronym: RESPONSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Philipp S. Muether, MD, PhD, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESPONSE2010
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab as needed (Other)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — upload (three monthly injections), re-treatment as needed
  Other Names: Lucentis

SUMMARY:
To assess genetic features and intraocular cytokine profiles of non-responders to anti-VEGF treatment of exudative age-related macular degeneration. Also to assess necessity and frequency of pro re nate medical re-treatment.

ELIGIBILITY:
Inclusion Criteria:

* active subfoveal CNV related to exudative age-related macular degeneration (all subforms)
* age > 60 years
* visual acuity > 20/400
* no previous treatment for AMD

Exclusion Criteria:

* any previous AMD therapy
* other CNV types (myopic, parapapillary)
* contraindication for ranibizumab treatment
* prior study participation for AMD
* pregnancy / premenopausal women

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 2 years
  Change in visual acuity within the observation period

SECONDARY OUTCOMES:
Association between treatment response and genotype | 2 years
Changes in OCT central retinal thickness / retinal volume | 2 years
Association between treatment application delay and visual outcome | 2 years
Association between re-treatment necessity / frequency and intraocular cytokine profiles | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philipp S Muether, MD, Principal Investigator — Center of Ophthalmology, University of Cologne
Locations (1):
- University Center of Ophthalmology, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Fauser S, Muether PS. Clinical correlation to differences in ranibizumab and aflibercept vascular endothelial growth factor suppression times. Br J Ophthalmol. 2016 Nov;100(11):1494-1498. doi: 10.1136/bjophthalmol-2015-308264. Epub 2016 Feb 17. PMID 26888975
- [Derived] Saunders DJ, Muether PS, Fauser S. A model of the ocular pharmacokinetics involved in the therapy of neovascular age-related macular degeneration with ranibizumab. Br J Ophthalmol. 2015 Nov;99(11):1554-9. doi: 10.1136/bjophthalmol-2015-306771. Epub 2015 May 8. PMID 25957377
- [Derived] Koch KR, Muether PS, Hermann MM, Hoerster R, Kirchhof B, Fauser S. Subjective perception versus objective outcome after intravitreal ranibizumab for exudative AMD. Graefes Arch Clin Exp Ophthalmol. 2012 Feb;250(2):201-9. doi: 10.1007/s00417-011-1792-8. Epub 2011 Sep 8. PMID 21901296